CLINICAL TRIAL: NCT02327650
Title: The Examinations Whether or Not the Primary Causes of Osteoarthritis or Rheumatoid Arthritis in Joints Might be Bone Alterations
Brief Title: To Examine Whether or Not the Primary Causes of OA or RA Might be Bone Alterations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant Professor, Shinshu University
Other Study IDs: OA RA Bone Study
Record Dates: First submitted 2014-12-21; First posted 2014-12-30 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Progression of Rheumatoid Arthritis; Osteoarthritis of Multiple Joints

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RA and OA: Every 2 or 3 months, plain radiograph, blood and urinary tests, and MRI are performed in the painful joints of RA.
  Interventions: Procedure: The examinations for bones in joints of OA and RA patients

INTERVENTIONS:
Procedure: The examinations for bones in joints of OA and RA patients

SUMMARY:
Generally, osteoarthris (OA) is considered as primarily cartilage disease. However, as we and others have previously reported, a portion of OA might be caused primarily by bone alterations. In this study, we prospectively and retrospectively show that the bone altertations may affect OA primarily in all of the joints.

In addition, rheumatoid arthritis (RA) is a joint disease when immune system attacks synovium. Joint destruction occurrs continuously if suitable treatment is not performed. The etiology of RA is still largely unknown. As with OA, RA can be primarily damaged in bone, instead of cartilage. Here we prospectively and retrospectively show that the bone altertations may affect RA primarily in all of the joints.

ELIGIBILITY:
Inclusion Criteria:

* RA and/or OA

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients who have OA with accompaying joint pain or the patients who have RA with accompaying joint pain
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The bone signal changes detected by MRI in OA and/or RA patients | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Yukio Nakamura, Matsumoto, Nagano
  - Yukio Nakamura, Matsumoto